CLINICAL TRIAL: NCT06163599
Title: Reducing Mental Health Disparities Among Latinxs With a Telenovela Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1864886-2
Record Dates: First submitted 2023-11-22; First posted 2023-12-11 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Anxiety Disorders
Keywords: anxiety disorder; transdiagnostic Treatment; United Protocol
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telenovela Arm (Experimental): The UP telenovela (which is the experimental treatment arm) constitutes of nine videos depicting the main character, Esperanza, who is struggling with anxiety and depression, undergoing therapy involving the UP, and completing worksheets relating to the weekly therapy sessions.
  Interventions: Behavioral: Transdiagnostic Telenovela Intervention

INTERVENTIONS:
Behavioral: Transdiagnostic Telenovela Intervention — The intervention constitutes nine videos depicting the main character, Esperanza, who is struggling with anxiety and depression, undergoing therapy involving the a trandiagnostic treatment, and completing worksheets relating to the weekly therapy sessions.

SUMMARY:
The primary aim of our study is to determine the effectiveness of an transdiagnostic telenovela video intervention in reducing anxiety and depressive symptoms using a pre/post-test design with Spanish-speaking Latinxs.

DETAILED DESCRIPTION:
Telenovela video interventions are a low-resource, low-cost methodology developed to diminish the treatment-provider gap (Heilemann et al., 2017). Research shows that telenovela interventions represent an acceptable (Heilemann et al., 2018) and potent (Heilemann et al., 2017) intervention option for disseminating information to the Latinx population. Prior research utilizing transmedia telenovela interventions that include a telenovela component have demonstrated some effectiveness at reducing symptoms of anxiety and depression among Latinxs (Heilemann et al., 2017; Kajiyama et al., 2018) as have fotonovelas (Sanchez et al., 2019). To date researchers have not investigated how the telenovela approach combined with a transdiagnostic treatment paradigm might help reduce behavioral health disparities among Spanish-speaking Latinxs given that such an intervention would be easily disseminable and target the two most common disorders observed among this population. The primary aim of this study is to determine the effectiveness of an transdiagnostic telenovela video intervention in reducing anxiety and depressive symptoms using a pre/post-test design with Spanish-speaking Latinxs.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Identify as Latinx
3. Prefer behavioral health services in Spanish
4. Meet the DSM criteria for any mild to moderate anxiety disorder
5. Ownership of a smartphone

Exclusion Criteria:

1. Suicidality
2. Psychosis
3. Bipolar disorder
4. Severe anxiety disorders
5. Severe depressive disorders
6. Homicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 | Two weeks
  Assesses the presence of anxiety symptoms in the past two weeks. Lower scores mean better outcomes. Scores range from 0 to 35.

CONTACTS AND LOCATIONS:
Locations (1):
- La Clinica @ the UNR Psychological Services Center, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided